CLINICAL TRIAL: NCT02527902
Title: Autonomic Nervous System (ANS) Analysis According to Different Renal Function Stage in Immunoglobin A (IgA) Nephropathy
Brief Title: Autonomic Nervous System (ANS) and Renal Function in Immunoglobin A (IgA) Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1008123
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: IGA Glomerulonephritis
Keywords: IGA Glomerulonephritis; Autonomic nervous system; ANS
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- IgAN with glomerular filtration rate (GFR) >90 ml/min/1.73 m2 (Experimental): Measure of ANS by holter device in IgAN patients with glomerular filtration rate (GFR) >90 ml/min/1.73 m2
  Interventions: Device: Holter
- IgAN with GFR 60-89 ml/min/1.73 m2 (Experimental): Measure of ANS by holter device in IgAN patients with GFR 60-89 ml/min/1.73 m2
  Interventions: Device: Holter
- IgAN with GFR 30-59 ml/min/1.73 m2 (Experimental): Measure of ANS by holter device in IgAN patients with GFR 30-59 ml/min/1.73 m2
  Interventions: Device: Holter
- IgAN with GFR 15-29 ml/min/1.73 m2 (Experimental): Measure of ANS by holter device in IgAN patients with GFR 15-29 ml/min/1.73 m2
  Interventions: Device: Holter
- IgAN with GFR < 15ml/min/1.73 m2 (Experimental): Measure of ANS by holter device in IgAN patients with GFR < 15ml/min/1.73 m2.
  Interventions: Device: Holter

INTERVENTIONS:
Device: Holter — measure of ANS in IgAN patients

SUMMARY:
The estimation of the cardiovascular risk in the general population must take into account small renal disturbances, as the microalbuminuria. Conversely certain parameters of the cardiovascular risk influence the evolution of renal diseases, for example the arterial high blood pressure.

The measure of the activity of the autonomous nervous system, and especially the quantification of its variability, is a means to estimate the cardiovascular risk. The investigators formulate the hypothesis that the variability of the autonomous nervous system is an additional clinical element for the evaluation of the evolutionary risk of renal diseases.

The aim of this study is to compare the variability of the autonomous nervous system during the various evolutionary stages of the renal disease.

The renal disease studied will be IgA nephropathy (IgNA). IgNA is a histologically defined glomerulonephritis (rela biopsy) by the presence of deposits immunoglobulin A (IgA) in the renal mesangium (at list 1+) by immunofluorescence.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of IgNA biopsy-proven free, informed, express and written

Exclusion Criteria:

* IgNA secondary to Henoch-Schonlein purpura (HSP) or Systemic Lupus Erythematosus or alcoholic cirrhosis
* current kidney transplantation
* Hypertension treated or not,
* Diseases interfering with ANS analysis: cardiac arrhythmia, beta-blocker therapy
* diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Standard deviation of all R-R intervals (SDNN) | day 1
  Comparison of Standard deviation of all R-R intervals (SDNN) between GFR category of IgNA

CONTACTS AND LOCATIONS:
Overall Officials: Eric Alamartine, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France